CLINICAL TRIAL: NCT05835739
Title: InheriteD brEast caNcer iTalian regIsTrY A Retrospective-prospective Observational Cohort Study to Evaluate Cancer Prevention Strategies in Women With a Deleterious Mutation in BRCA1-2
Acronym: IDENTITY
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2019-33
Record Dates: First submitted 2023-03-24; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (Retrospective): all consecutive women with a germline deleterious mutation in BRCA1-2 admitted to the participant Center since 1st of January 2010 until site activation will be enrolled
- Cohort B (Prospective):: all consecutive women with a germline deleterious mutation in BRCA1-2 admitted to the participant Center since site activation until September 2025 will be enrolled

SUMMARY:
The purpose of the study is to obtain and centralize data about cancer prevention strategies in women with a germline deleterious mutation in BRCA1-2 with or without a history of breast cancer in Italy

DETAILED DESCRIPTION:
Women who carry a deleterious mutation in breast cancer susceptibility gene 1 (BRCA1) or breast cancer susceptibility gene 2 (BRCA2) have an elevated lifetime risk of developing breast and ovarian cancer, estimated at up to 7 and 25 times that of the average risk population, respectively. By the age of 80 years, the estimated cumulative risk of breast cancer is about 70% for BRCA1/2 mutation carriers, while the cumulative ovarian cancer risk is about 40% for BRCA1 and 20% for BRCA2 carriers. Thus, BRCA1/2 mutation carriers are advised to consider different risk-reducing strategies, including surveillance (breast self-examination, clinical breast examination, screening using mammography, ultrasound and breast magnetic resonance imaging), chemoprevention and prophylactic surgery (prophylactic mastectomy and/or salpingo-oophorectomy). Prospective cohort studies demonstrate that risk-reducing mastectomy is associated with 90% or more decreased risk of breast cancer. Unfortunately, it is difficult to quantify its effect on overall mortality since no randomized studies have compared risk-reducing mastectomy with enhanced screening, risk-reducing salpingo oophorectomy or prophylactic treatment. Additionally, prophylactic mastectomy is an invasive intervention associated with a substantial complication rate and psychological distress, changes in body image and sexual function. Therefore, as a preventive measure, risk-reducing mastectomy should be discussed on a case-by case basis, after proper counseling regarding benefits, limitations, risks of surgical complications and psychosocial impact. Conversely, risk-reducing salpingo oophorectomy is strongly recommended for women with mutations in BRCA1 (between ages 35 and 40 years) and BRCA2 (between ages 40 and 45 years) after completion of childbearing desire, for a significant reduction in ovarian cancer incidence and all-cause mortality. In the absence of solid evidences coming from randomized clinical trials, the aim of the present study is to collect and centralize real-world data on cancer prevention strategies (prophylactic surgery, prophylactic therapies, active surveillance) and oncologic treatments of women with a deleterious mutation in BRCA1-2 with or without a diagnosis of breast cancer in Italy. By collecting and analyzing these data, the IDENTITY study aims to obtain a faithful representation of the practices related to oncological surveillance in the group of patients analyzed.

ELIGIBILITY:
Inclusion Criteria:

Cohort A (Retrospective):

1. Female sex
2. Age ≥ 18 years
3. Signed informed consent
4. Documented germline deleterious mutation in BRCA1 and/or BRCA2 in people with: i) No history of cancer ii) Radically treated breast cancer iii) Stage IV breast cancer diagnosed after BRCA1-2 mutation detection
5. Admission to the participating Center since 1st of January 2010, prior to site activation

Cohort B (Prospective):

1. Female sex
2. Age ≥ 18 years
3. Signed informed consent
4. Documented germline deleterious mutation in BRCA1 and/or BRCA2 in people with: i) No history of cancer ii) Radically treated breast cancer iii) Stage IV breast cancer diagnosed after BRCA1-2 mutation detection
5. Admission to the participating Center after site activation

Exclusion Criteria:

Cohort A/B (Retrospective/Prospective):

1. Other malignancies diagnosed within five years prior to BRCA1-2 mutation detection, except for:

* ovarian cancer stage I-II
* basal or squamous cell carcinoma of the skin
* melanoma in situ
* CIS of the cervix

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV breast cancer diagnosed after BRCA1-2 mutation detection
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2035-09-30 (Estimated)

PRIMARY OUTCOMES:
To obtain and centralize data about cancer prevention strategies in women with a germline deleterious mutation in BRCA1-2 with or without a history of breast cancer in Italy | 10 years since enrolment
  To obtain and centralize data about cancer prevention strategies in women with a germline deleterious mutation in BRCA1-2 with or without a history of breast cancer in Italy

SECONDARY OUTCOMES:
To evaluate the clinico-radiological follow-up (type and frequency) of women with a germline deleterious mutation in BRCA1-2 with or without a history of early breast cancer | 10 years since enrolment
  To evaluate the clinico-radiological follow-up (type and frequency) of women with a germline deleterious mutation in BRCA1-2 with or without a history of early breast cancer
To evaluate the treatment of early and/or advanced breast cancer in women with a germline deleterious mutation in BRCA1-2 | 10 years since enrolment
  To evaluate the treatment of early and/or advanced breast cancer in women with a germline deleterious mutation in BRCA1-2
To evaluate disease-free survival and/or progression-free survival and overall survival of women with a germline deleterious mutation in BRCA1-2 treated for early and/or advanced breast cancer | 10 years since enrolment
  To evaluate disease-free survival and/or progression-free survival and overall survival of women with a germline deleterious mutation in BRCA1-2 treated for early and/or advanced breast cancer

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - Centro di Riferimento Oncologico - Aviano, Aviano, Pordenone
  - IRCCS AOU San Martino, IST Genova, Genova
  - Azienda Ospedaliera Papardo, Messina
  - ASST Ovest Milanese, Milan
  - Azienda ospedaliera Universitaria di Modena, Modena
  - Università degli studi di Napoli Federico II, Napoli
  - Azienda AUSL IRCCS - Reggio Emilia, Reggio Emilia
  - ASL Roma 1, Santo Spirito, Roma
  - IFO - Istituto Regina Elena (Oncologia medica 2), Roma
  - Policlinico Universitario Gemelli, Roma
  - Città della salute Torino, PO S. Anna, Torino
  - ASU FC Azienda Sanitaria Universitaria Friuli Centrale, Udine

REFERENCES:
- [Result] Paul A, Paul S. The breast cancer susceptibility genes (BRCA) in breast and ovarian cancers. Front Biosci (Landmark Ed). 2014 Jan 1;19(4):605-18. doi: 10.2741/4230. PMID 24389207
- [Result] King MC, Marks JH, Mandell JB; New York Breast Cancer Study Group. Breast and ovarian cancer risks due to inherited mutations in BRCA1 and BRCA2. Science. 2003 Oct 24;302(5645):643-6. doi: 10.1126/science.1088759. PMID 14576434
- [Result] Kuchenbaecker KB, Hopper JL, Barnes DR, Phillips KA, Mooij TM, Roos-Blom MJ, Jervis S, van Leeuwen FE, Milne RL, Andrieu N, Goldgar DE, Terry MB, Rookus MA, Easton DF, Antoniou AC; BRCA1 and BRCA2 Cohort Consortium; McGuffog L, Evans DG, Barrowdale D, Frost D, Adlard J, Ong KR, Izatt L, Tischkowitz M, Eeles R, Davidson R, Hodgson S, Ellis S, Nogues C, Lasset C, Stoppa-Lyonnet D, Fricker JP, Faivre L, Berthet P, Hooning MJ, van der Kolk LE, Kets CM, Adank MA, John EM, Chung WK, Andrulis IL, Southey M, Daly MB, Buys SS, Osorio A, Engel C, Kast K, Schmutzler RK, Caldes T, Jakubowska A, Simard J, Friedlander ML, McLachlan SA, Machackova E, Foretova L, Tan YY, Singer CF, Olah E, Gerdes AM, Arver B, Olsson H. Risks of Breast, Ovarian, and Contralateral Breast Cancer for BRCA1 and BRCA2 Mutation Carriers. JAMA. 2017 Jun 20;317(23):2402-2416. doi: 10.1001/jama.2017.7112. PMID 28632866
- [Result] Rebbeck TR, Mitra N, Wan F, Sinilnikova OM, Healey S, McGuffog L, Mazoyer S, Chenevix-Trench G, Easton DF, Antoniou AC, Nathanson KL; CIMBA Consortium; Laitman Y, Kushnir A, Paluch-Shimon S, Berger R, Zidan J, Friedman E, Ehrencrona H, Stenmark-Askmalm M, Einbeigi Z, Loman N, Harbst K, Rantala J, Melin B, Huo D, Olopade OI, Seldon J, Ganz PA, Nussbaum RL, Chan SB, Odunsi K, Gayther SA, Domchek SM, Arun BK, Lu KH, Mitchell G, Karlan BY, Walsh C, Lester J, Godwin AK, Pathak H, Ross E, Daly MB, Whittemore AS, John EM, Miron A, Terry MB, Chung WK, Goldgar DE, Buys SS, Janavicius R, Tihomirova L, Tung N, Dorfling CM, van Rensburg EJ, Steele L, Neuhausen SL, Ding YC, Ejlertsen B, Gerdes AM, Hansen Tv, Ramon y Cajal T, Osorio A, Benitez J, Godino J, Tejada MI, Duran M, Weitzel JN, Bobolis KA, Sand SR, Fontaine A, Savarese A, Pasini B, Peissel B, Bonanni B, Zaffaroni D, Vignolo-Lutati F, Scuvera G, Giannini G, Bernard L, Genuardi M, Radice P, Dolcetti R, Manoukian S, Pensotti V, Gismondi V, Yannoukakos D, Fostira F, Garber J, Torres D, Rashid MU, Hamann U, Peock S, Frost D, Platte R, Evans DG, Eeles R, Davidson R, Eccles D, Cole T, Cook J, Brewer C, Hodgson S, Morrison PJ, Walker L, Porteous ME, Kennedy MJ, Izatt L, Adlard J, Donaldson A, Ellis S, Sharma P, Schmutzler RK, Wappenschmidt B, Becker A, Rhiem K, Hahnen E, Engel C, Meindl A, Engert S, Ditsch N, Arnold N, Plendl HJ, Mundhenke C, Niederacher D, Fleisch M, Sutter C, Bartram CR, Dikow N, Wang-Gohrke S, Gadzicki D, Steinemann D, Kast K, Beer M, Varon-Mateeva R, Gehrig A, Weber BH, Stoppa-Lyonnet D, Sinilnikova OM, Mazoyer S, Houdayer C, Belotti M, Gauthier-Villars M, Damiola F, Boutry-Kryza N, Lasset C, Sobol H, Peyrat JP, Muller D, Fricker JP, Collonge-Rame MA, Mortemousque I, Nogues C, Rouleau E, Isaacs C, De Paepe A, Poppe B, Claes K, De Leeneer K, Piedmonte M, Rodriguez G, Wakely K, Boggess J, Blank SV, Basil J, Azodi M, Phillips KA, Caldes T, de la Hoya M, Romero A, Nevanlinna H, Aittomaki K, van der Hout AH, Hogervorst FB, Verhoef S, Collee JM, Seynaeve C, Oosterwijk JC, Gille JJ, Wijnen JT, Gomez Garcia EB, Kets CM, Ausems MG, Aalfs CM, Devilee P, Mensenkamp AR, Kwong A, Olah E, Papp J, Diez O, Lazaro C, Darder E, Blanco I, Salinas M, Jakubowska A, Lubinski J, Gronwald J, Jaworska-Bieniek K, Durda K, Sukiennicki G, Huzarski T, Byrski T, Cybulski C, Toloczko-Grabarek A, Zlowocka-Perlowska E, Menkiszak J, Arason A, Barkardottir RB, Simard J, Laframboise R, Montagna M, Agata S, Alducci E, Peixoto A, Teixeira MR, Spurdle AB, Lee MH, Park SK, Kim SW, Friebel TM, Couch FJ, Lindor NM, Pankratz VS, Guidugli L, Wang X, Tischkowitz M, Foretova L, Vijai J, Offit K, Robson M, Rau-Murthy R, Kauff N, Fink-Retter A, Singer CF, Rappaport C, Gschwantler-Kaulich D, Pfeiler G, Tea MK, Berger A, Greene MH, Mai PL, Imyanitov EN, Toland AE, Senter L, Bojesen A, Pedersen IS, Skytte AB, Sunde L, Thomassen M, Moeller ST, Kruse TA, Jensen UB, Caligo MA, Aretini P, Teo SH, Selkirk CG, Hulick PJ, Andrulis I. Association of type and location of BRCA1 and BRCA2 mutations with risk of breast and ovarian cancer. JAMA. 2015 Apr 7;313(13):1347-61. doi: 10.1001/jama.2014.5985. PMID 25849179
- [Result] Carbine NE, Lostumbo L, Wallace J, Ko H. Risk-reducing mastectomy for the prevention of primary breast cancer. Cochrane Database Syst Rev. 2018 Apr 5;4(4):CD002748. doi: 10.1002/14651858.CD002748.pub4. PMID 29620792
- [Result] Heemskerk-Gerritsen BA, Menke-Pluijmers MB, Jager A, Tilanus-Linthorst MM, Koppert LB, Obdeijn IM, van Deurzen CH, Collee JM, Seynaeve C, Hooning MJ. Substantial breast cancer risk reduction and potential survival benefit after bilateral mastectomy when compared with surveillance in healthy BRCA1 and BRCA2 mutation carriers: a prospective analysis. Ann Oncol. 2013 Aug;24(8):2029-35. doi: 10.1093/annonc/mdt134. Epub 2013 Apr 10. PMID 23576707